CLINICAL TRIAL: NCT01421810
Title: Ovarian Contribution to Androgen Production in Adolescent Girls
Acronym: CBS001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Christine Burt Solorzano, Assistant Professor in Pediatrics, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15298
Record Dates: First submitted 2011-08-17; First posted 2011-08-23 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Polycystic Ovary Syndrome; Obesity; Hyperandrogenism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity; Hyperandrogenism | interventions — Dexamethasone; Ovidrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dexamethasone, rhCG (Ovidrel) (Experimental): rhCG (Ovidrel) administered 25 mcg IV; dexamethasone administered 1 mg PO
  Interventions: Drug: Dexamethasone; Drug: rhCG

INTERVENTIONS:
Drug: Dexamethasone — 1 mg PO
Drug: rhCG — 25 mcg IV
  Other Names: (Ovidrel)

SUMMARY:
Women with polycystic ovary syndrome (PCOS) can have unwanted facial or male-patterned body hair, irregular menstrual periods, or no menstrual periods excess body weight, and infertility. It also results in elevated androgen levels such as testosterone. In women with PCOS, the majority of excess androgens are produced by the ovaries. However, it is unknown whether the ovaries are fully active during early puberty. The purpose of this study is to determine how the ovaries contribute to the production of male hormones in the body during different stages of puberty, so that it can be better understood why some females have excess androgens.

DETAILED DESCRIPTION:
Adolescent hyperandrogenemia can represent a forerunner to adult PCOS. Because adrenarche leads to an increase in adrenal androgen production during early puberty and since early puberty is associated with an overnight rise in testosterone that follows a similar time course to cortisol, we hypothesize that the adrenal gland is a major source of androgens in early puberty. On the other hand, the overnight rise in testosterone may reflect an ovarian response to overnight increases of gonadotropin secretion in early puberty. However, the ability of the ovaries to produce androgens (e.g., to respond to gonadotropin stimulation) during early puberty has not been tested concurrently in these girls. The sources of excess androgen production and the timing of their relative contributions across puberty are important in understanding the mechanism of hyperandrogenemia in these individuals. In addition, determination of the sources of hyperandrogenemia across puberty may have clinical utility in the development of preclinical screening tests designed to reveal those girls at greatest risk for PCOS and identification of potential therapeutic targets to prevent its development.

ELIGIBILITY:
Inclusion Criteria:

* Girls age 7-18 years
* Normal weight (BMI 5-85%-ile for age) or overweight (>85%-ile)
* With or without signs of excess androgen
* Screening labs within age-appropriate normal range, with the exception of a mildly low hematocrit (see below) and the hormonal abnormalities inherent in obesity which could include mildly elevated luteinizing hormone (LH), lipids, testosterone, prolactin, DHEAS, E2, glucose, and insulin; and decreased follicle-stimulating hormone (FSH) and/or sex hormone-binding globulin (SHBG)

Exclusion Criteria:

* Patients currently enrolled in another research protocol will be excluded, except for those enrolled in IRB-HSR #12702/JCM022. This protocol is designed to allow subjects enrolling in IRB-HSR #12702/JCM022 to simultaneously participate in this companion protocol.
* Inability to comprehend what will be done during the study or why it will be done
* BMI-for-age < 5th percentile
* Weight < 27 kg if simultaneously participating in IRB-HSR #12702/JCM022 due to blood volume limits
* Obesity associated with a diagnosed genetic syndrome (e.g. Prader-Willi syndrome)
* Since the study involves looking at ovarian function, boys will be excluded.
* Positive pregnancy test or lactation. Subjects with a positive pregnancy test will be informed of the result by the screening physician. Under Virginia law, parental notification is not required for minors. However, the screening physician will encourage them to tell their parent(s) and counsel them about the importance of appropriate prenatal care and counseling. We will arrange follow-up for them at the Teen Health Clinic at the University of Virginia or their primary care physician's office in a timely manner.
* Abnormal laboratory studies will be confirmed by repeat testing to exclude laboratory error.
* Morning cortisol < 3 microgram/dL or history of Cushing syndrome or adrenal insufficiency
* History of congenital adrenal hyperplasia or 17-hydroxyprogesterone > 300 ng/dL, which suggests the possibility of congenital adrenal hyperplasia (if postmenarchal, the 17-hydroxyprogesterone will be collected during the follicular phase, or ≥ 40 days since last menses if oligomenorrheic). NOTE: If a 17-hydroxyprogesterone >300 mg/dL is confirmed on repeat testing, an adrenocorticotropic hormone-stimulated 17-hydroxyprogesterone <1000 ng/dL will be required for study participation.
* Total testosterone > 150 ng/dL
* Previous diagnosis of diabetes, fasting glucose ≥126 mg/dL, or a hemoglobin A1c >6.5%
* Abnormal thyroid stimulating hormone (TSH) for age. Subjects with adequately treated hypothyroidism, reflected by normal TSH values, will not be excluded.
* Abnormal prolactin. Mild elevations may be seen in overweight girls, and elevations <1.5 times the upper limit of normal will be accepted in this group.
* Persistent hematocrit <36% and hemoglobin <12 g/dL. Subjects with a mildly low hematocrit (33-36%) will be asked to take iron in the form of ferrous gluconate for up to 60 days. Subjects weighing ≤ 36 kg will take one 300-325 mg tablet oral ferrous gluconate daily (containing 36 mg elemental iron); subjects weighing >36 kg will take two 300-325 mg tablets oral ferrous gluconate daily (containing 36 mg elemental iron each). They will return to the Clinical Research Unit (CRU) or alternate UVA clinical unit after 30-60 days of iron therapy to have their hemoglobin or hematocrit rechecked and will proceed with the remainder of the study if it is ≥12 g/dL or ≥36%, respectively.
* Persistent liver test abnormalities, with the exception that mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome. Mild elevations may be seen in overweight girls, so elevations <1.5 times the upper limit of normal will be accepted in this group.

Ages: 7 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-03-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assess baseline and stimulated ovarian hormone levels in response to recombinant human chorionic gonadotropin (rhCG) administration in normal weight and overweight girls across puberty | 24 hours after administration of rhCG administration

CONTACTS AND LOCATIONS:
Overall Officials: Christine Burt Solorzano, MD, Principal Investigator — University of Virginia Center for Research in Reproduction
Locations (1):
- University of Virginia Center for Research in Reproduction, Charlottesville, Virginia, United States